CLINICAL TRIAL: NCT03426787
Title: Development and Validation of a Shared-decision Making Tool for Initiation of Treatment in Patients With Hepatitis C Infection and Advanced Chronic Kidney Disease
Brief Title: Helping Empower Liver and Kidney Patients
Acronym: Project HELP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Mary C. Politi, Associate Professor of Surgery, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201707154
Record Dates: First submitted 2018-01-21; First posted 2018-02-08 (Actual); Results first posted 2019-07-05 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Hepatitis C; Chronic Kidney Diseases; Patient Education
Keywords: Patient Centered; Pre-Post Design; Decision Support; Health Literacy
MeSH Terms: conditions — Hepatitis C; Renal Insufficiency, Chronic | interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: pre-post within subjects design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Aid (Experimental): A decision supports tool that guides patients with Hepatitis C and Chronic Kidney Disease through choices about whether, when, and how to treat each illness.
  Interventions: Behavioral: Decision Aid

INTERVENTIONS:
Behavioral: Decision Aid — Participants will have the option to view a web or paper-based version of the decision aid.

SUMMARY:
The overall purpose of this study is to develop and test a web-based decision aid (DA) to support patients with Hepatitis C and Chronic Kidney Disease during decisions about whether, when, and how to treat each illness. Patients will have the opportunity to learn about their hepatitis C and kidney disease, initiate thought about what matters most to them and choose a treatment plan for their liver and kidney disease that works best for them. Investigators will evaluate the tool's efficacy, usability, and the likelihood of using it in clinical practice. There are three (3) primary aims of this project: (1) to develop the DA; (2) to pilot-test the DA to determine efficacy, usability and likelihood of using it in routine practice; (3) to explore stakeholders feedback on the usefulness of the DA and likelihood of implementing the tool.

DETAILED DESCRIPTION:
First, for Aim 1, Investigators along with direction from a diverse expert advisory group of nephrologists, hepatologists, and patient partners developed a decision aid based upon International Patient Decision Aids Standards guidelines, literature reviews, and expert advisory reviews. It includes plain language education, interactive learning modules personalized tailored information to help individuals use and consider information appropriate to their values and needs, and guidance on discussions with clinicians about treatment goals. Second, for Aim 2, Investigators will pilot-test the decision aid with 70 individuals in a pre-post within-subjects study design to evaluate the tool's efficacy, usability, and the likelihood of using it in clinical practice. Lastly, for Aim 3, Investigators will conduct 30 semi-structured qualitative interviews with both clinicians and participants after the pilot evaluation of the decision aid to gather feedback about implementing the tool into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Must read and understand English AND
* Must have Hepatitis C (any genotype) and Chronic Kidney Disease (any stage)

Exclusion Criteria:

* Developed jaundice, ascites, variceal hemorrhage, or hepatic encephalopathy also known as Decompensated cirrhosis; or
* Currently has or had liver cancer (Hepatocellular carcinoma); or
* Received a liver transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2019-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Politi, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] George N, Liapakis A, Korenblat KM, Li T, Roth D, Yee J, Fowler KJ, Howard L, Liu J, Politi MC. A Patient Decision Support Tool for Hepatitis C Virus and CKD Treatment. Kidney Med. 2019 Jul 11;1(4):200-206. doi: 10.1016/j.xkme.2019.06.003. eCollection 2019 Jul-Aug. PMID 32734200
- See also: Decisional Conflict Scale Measure — https://decisionaid.ohri.ca/eval_dcs.html
- See also: Decision Self-Efficacy Scale Measure — https://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Decision_SelfEfficacy.pdf
- See also: Usability Scale Measure — https://www.usability.gov/how-to-and-tools/methods/system-usability-scale.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Project HELP Decision Aid: A decision supports tool that guides patients with Hepatitis C and Chronic Kidney Disease through choices about whether, when, and how to treat each illness. Participants will have the option to view a web or paper-based version of the decision aid.
Period: Overall Study
Arm/Group | Project HELP Decision Aid
Started | 70
Completed | 56
Not Completed | 14
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 7
Not completed — Unrelated to intervention death | 1

BASELINE CHARACTERISTICS:
Groups:
- Decision Support Tool: A decision supports tool that guides patients with Hepatitis C and Chronic Kidney Disease through choices about whether, when, and how to treat each illness.
  Decision Aid: Participants will have the option to view a web or paper-based version of the decision aid.
Arm/Group | Decision Support Tool
Number analyzed (Participants) | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.95 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 46
  White | 7
  More than one race | 2
  Unknown or Not Reported | 0
Education [Count of Participants; unit: Participants]
  Less than or some high school | 22
  High school diploma or GED | 13
  Technical Training or Certification | 5
  Some college | 11
  College degree or highe | 5
Type of Insurance Coverage [Count of Participants; unit: Participants]
  Private | 2
  Governmental (Medicaid, Medicare, & VA/TriCare | 52
  Uninsured | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Knowledge
Description: The percent correct out of eight questions created by the research team based on information that is considered vital to making treatment decisions, including understanding HCV and CKD, the health effects of both diseases, and understanding factors that differentiate treatment options. Scores range from 0 to 100. Higher scores demonstrate more knowledge.
Time Frame: At baseline and immediately after viewing the intervention, within 30 minutes.
Population: Participants completed both pre and post-test survey questions for the knowledge questions.
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Groups:
- Knowledge Pre-Test Scores: Participants knowledge scores at the baseline level.
- Knowledge Post Test Scores: Participants knowledge scores after using intervention
Arm/Group | Knowledge Pre-Test Scores | Knowledge Post Test Scores
Number analyzed (Participants) | 56 | 54
percentage of correct responses | 53.54 (21.31) | 65.74 (22.80)
Statistical Analysis 1: Comparison: Knowledge Pre-Test Scores vs Knowledge Post Test Scores; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -12.30216, 95% CI 2-sided [-18.95 to -5.6531]

2. Primary Outcome: Change in Decisional Conflict Scale
Description: The validated, 4-item SURE Test for clinical practice will be used. This scale measures whether individuals feel they have enough information to make a choice, are clear about their values for risks and benefits of their choice and feel they have enough support to make a choice. Scores range from 0 to 4. Higher scores indicate more confidence in their choice.
Time Frame: At baseline and immediately after viewing the intervention, within 30 minutes.
Population: Participants completed both pre and post-test survey questions for the decisional conflict scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Decisional Conflict Pre-Test Scores: Participants knowledge scores at the baseline level.
- Decisional Conflict Post Test Scores: Participants knowledge scores after using intervention
Arm/Group | Decisional Conflict Pre-Test Scores | Decisional Conflict Post Test Scores
Number analyzed (Participants) | 55 | 54
score on a scale | 2.64 (1.38) | 3.13 (1.40)
Statistical Analysis 1: Comparison: Decisional Conflict Pre-Test Scores vs Decisional Conflict Post Test Scores; Test type: Superiority; p = 0.0463, t-test, 2 sided; Mean Difference (Final Values) = -0.4717, 95% CI 2-sided [-0.9355 to -0.00793]

3. Primary Outcome: Change in Decision Self-Efficacy Scale
Description: The validated decision self-efficacy scale will be used. This 11-item scale measures an individual's self-confidence or belief in their ability to make a decision. Individuals will be asked to rate how confident they feel taking actions involved in making an informed choice (e.g., gathering information, asking questions, and expressing opinions). Scores can range from 0 to 100. Higher scores indicate more confidence in participants ability to make a treatment choice.
Time Frame: At baseline and immediately after viewing the intervention, within 30 minutes.
Population: Participants completed both pre and post-test survey questions for the decision self-efficacy scale.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Decision Self Efficacy Pre-Test Scores: Participants decision self-efficacy scores at the baseline level.
- Decision Self Efficacy Post Test Scores: Participants decision self-efficacy scores after using intervention
Arm/Group | Decision Self Efficacy Pre-Test Scores | Decision Self Efficacy Post Test Scores
Number analyzed (Participants) | 56 | 54
score on a scale | 84.42 (17.07) | 86.62 (18.88)
Statistical Analysis 1: Comparison: Decision Self Efficacy Pre-Test Scores vs Decision Self Efficacy Post Test Scores; Test type: Superiority; p > 0.05, t-test, 2 sided; Median Difference (Final Values) = -1.9360, 95% CI 2-sided [-7.4086 to 3.5365]

4. Secondary Outcome: System Usability Scale
Description: A 10-item scale that evaluates the website's usability level. Scores can range from 0 to 100. An average score of 68 is considered a usable/adequate tool per measure guidelines. Higher scores represent better usability level for the tool.
Time Frame: Completed immediately after viewing the intervention
Population: Participants completed the system usability scale in our post-test questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project HELP Decision Aid
Number analyzed (Participants) | 54
score on a scale | 69.86 (20.43)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Project HELP Decision Aid
All-Cause Mortality (participants affected / at risk) | 1/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 0/70

LIMITATIONS AND CAVEATS:
Given the small sample and pilot study design, the reported observations can be interpreted as preliminary results. This project was also a single site study. Results might not be generalizable across other regions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/87/NCT03426787/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/87/NCT03426787/Prot_SAP_001.pdf